CLINICAL TRIAL: NCT05010434
Title: Sintilimab and Bevacizumab Combined With Radiotherapy in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Sintilimab and Bevacizumab Combined With Radiotherapy for Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRRHCC
Record Dates: First submitted 2021-08-14; First posted 2021-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab and Bevacizumab Combined with Radiotherapy (Experimental)
  Interventions: Drug: Sintilimab and Bevacizumab Combined with Radiotherapy

INTERVENTIONS:
Drug: Sintilimab and Bevacizumab Combined with Radiotherapy — Before radiotherapy: Bevacizumab+Sintilizumab, Q3w, 2 cycles in total. Radiation therapy: 30-50Gy/10 fractions. After radiotherapy: Bevacizumab+Sintilizumab, Q3w until disease progression or toxicity is intolerable.

SUMMARY:
The purpose of this study is to investigate both the efficacy and safety of sintilimab combined with bevacizumab and radiotherapy in advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
3. Treatment-naïve primary HCC (consistent with the American Association for the Study of Liver Diseases 2018 Guideline on Liver Cancer Diagnosis (18)) or initial recurrent HCC after radical resection without any postoperative anti-cancer treatment;
4. At least one measurable lesion in the liver on the basis of modified Response Evaluation Criteria in Solid Tumors (mRECIST);
5. Presented with Cheng's type I/II/III PVTT;
6. Largest tumor size ≤ 10 cm, number of tumors ≤ 3, and remnant liver volume ≥ 50%;
7. Child-Pugh class A;
8. Adequate hematological, liver, renal function:

   1. hemoglobin concentration ≥ 90 g/L;
   2. neutrophil count ≥ 1.5×109/L;
   3. platelet count ≥ 60×109/L;
   4. AST and ALT ≤ 3×upper limit of normal (ULN)
   5. total bilirubin ≤ 1.5×ULN;
   6. serum creatinine ≤ 1.5×ULN;
   7. serum albumin concentration ≥ 30 g/L;
9. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Tumor invasion of the superior mesenteric vein or bile ducts;
2. Infiltrative HCC;
3. Allergic to research reagents;
4. With other malignancies within 5 years;
5. With poorly controlled hypertension;
6. A past medical history of hepatic decompensation, such as hepatic encephalopathy, refractory ascites, and esophageal or gastric variceal bleeding;
7. A history of autoimmune disease;
8. Active infection requiring systemic treatments;
9. Severe bleeding;
10. With diseases needing daily non-steroidal anti-inflammatory drug (NSAID) therapy;
11. With other severe comorbidities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
ORR (objective response rate) | through study completion, up to 2 year
  the proportion of patients who have a partial or complete response to therapy.

SECONDARY OUTCOMES:
PFS (progression-free survival) | through study completion, up to 2 year
  defined as the time from receiving treatment until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.
OS (overall survival) | through study completion, up to 2 year
  defined as the time from receiving treatment until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.
DCR (disease control rate) | through study completion, up to 2 year
  the proportion of patients whose tumors have shrunk or been stable for a certain period of time, including cases of complete response (CR), partial response (PR), or stable disease (SD).
LCR (local control rate) | through study completion, up to 2 year
  the percentage of lesions with absence of recurrence within the high-dose region （80% isodose volume）
Adverse effects | through study completion, up to 2 year
  Adverse effects of sintilimab and bevacizumab combined with radiotherapy,number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu M, Liu Z, Chen S, Luo Z, Tu J, Qiao L, Wu J, Fan W, Peng Z. Sintilimab plus bevacizumab combined with radiotherapy as first-line treatment for hepatocellular carcinoma with portal vein tumor thrombus: A multicenter, single-arm, phase 2 study. Hepatology. 2024 Oct 1;80(4):807-815. doi: 10.1097/HEP.0000000000000776. Epub 2024 Feb 15. PMID 38358542